CLINICAL TRIAL: NCT05587335
Title: Project Harmony 2.0: A Relationship Education Intervention for Couples
Brief Title: Project Harmony 2.0: Relationship Education for Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCFloirda
Record Dates: First submitted 2022-09-22; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Marital Relationship

STUDY DESIGN:
Intervention Model Description: In person and online arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In person (Experimental): Couples will be assigned into in person relationship intervention.
  Interventions: Behavioral: PREP
- Online (Experimental): Couples will be assigned into online relationship intervention.
  Interventions: Behavioral: OurRelationship

INTERVENTIONS:
Behavioral: PREP — Relationship intervention to improve communication and conflict resolution for couples
  Arms: In person
Behavioral: OurRelationship — Relationship intervention to improve communication and conflict resolution for couples
  Arms: Online

SUMMARY:
Project Harmony directly addresses prioritized areas identified by Administration of Children and Families, emphasizing healthy marriage promotion activities and career advancement opportunities for adults. Included in service provisions are elements of: [a] marriage and relationship education/skills, [b] marriage enhancement, [c] divorce reduction and [d] job and career advancement. The targeted service population for Project Harmony includes married/committed couples in the greater Orlando metro area.

DETAILED DESCRIPTION:
The primary program consists of 12 hours of relationship education. The investigators seek to conduct an impact evaluation utilizing a randomized control trial (RCT) to compare outcomes of couples enrolled in either face to face relationship education or web-based relationship education to assess the impact of program structure on outcomes. By offering both face to face and online versions of evidenced based curricula, the investigators are directly addressing requests from ongoing needs assessments of our targeted population. The project is designed for couples 18 years and older; all participants in the face-to-face group will receive the Prevention and Relationship Education Program (PREP) 8.0 + Career Pathways Program (CPP) curricula whereas couples in the online group will receive the OurRelationship Intervention + CPP curricula.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years older and be in a committed relationship, must attend with partners

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1800 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Revised Dyadic Adjustment Scale | 6 months
  The Revised Dyadic Adjustment Scale (RDAS) is a self report questionnaire that assesses seven dimensions of couple relationships. The RDAS includes only 14 items, ranging from 0 to 69 with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress. The cut-off score for the RDAS is 48 such that scores of 48 and above indicate non-distress and scores of 47 and below indicate marital/relationship distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No